CLINICAL TRIAL: NCT02040857
Title: A Phase 2 Pilot Feasibility Study of Palbociclib in Combination With Adjuvant Endocrine Therapy for Hormone Receptor Positive Invasive Breast Carcinoma
Brief Title: Palbociclib in Combination With Adjuvant Endocrine Therapy for Hormone Receptor Positive, HER2 Negative Invasive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Erica Mayer, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-559
Record Dates: First submitted 2014-01-13; First posted 2014-01-20 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Aromatase Inhibitors; Letrozole; Anastrozole; exemestane; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palbociclib With Adjuvant Endocrine Therapy (Experimental): * Palbociclib 125 mg PO qd 21 days on, 7 days off
  * Endocrine Therapy: Tamoxifen 20mg, Letrozole 2.5mg, Anastrozole 1mg, or Exemestane 25mg PO qd
  Interventions: Drug: Palbociclib; Drug: Aromatase Inhibitor

INTERVENTIONS:
Drug: Palbociclib — CDK 4/6 inhibitor
  Other Names: PD 0332991-0054; PD-0332991; PD-332991; PF-00080665-73
Drug: Aromatase Inhibitor — Endocrine Therapy
  Other Names: Femara; Letrozole; Anastrozole; Arimidex; Exemestane; Aromasin; Tamoxifen; Nolvadex

SUMMARY:
This research study is evaluating a drug called Palbociclib in combination with endocrine therapy as a possible treatment for hormone receptor positive breast cancer.

* Palbociclib is a drug that may stop cancer cells from growing. Palbociclib blocks activity of two closely related enzymes (proteins that help chemical reactions in the body occur), called Cyclin D Kinases 4 and 6 (CDK 4/6). These proteins are part of a pathway, or a sequence of steps which is known to regulate cell growth. Laboratory testing has suggested palbociclib may stop the growth of hormone receptor positive breast cancer.
* Endocrine therapy prevents breast cancer cell growth by blocking estrogen stimulation. During this study endocrine therapy will either be tamoxifen or an aromatase inhibitor. It is standard of care for premenopausal women to take tamoxifen and for postmenopausal women to take either an aromatase inhibitor or tamoxifen after a diagnosis of hormone receptor positive breast cancer.

DETAILED DESCRIPTION:
After the screening procedures confirms that the participant is able to participate in the study. The participant will be given a dosing diary for each treatment cycle. Each treatment cycle lasts 28 days, during which time the participant will take Palbociclib once a day on days 1-21 of each 28 day cycle and the aromatase inhibitor that the participant is already taking once a day every day. The diary will also include special instructions for taking the study drug(s).

All participants participating in the research study will receive the same dose of Palbociclib.

While participating in the research study the participant will have the following tests and procedures:

* Clinical Exams: The participant will have a physical exam on the first day of the month for first three months of therapy. After that, the participant will have a physical exam every other month until the end of the first year of therapy. After the first year, the participant will have a physical exam every 3 months during the second year of therapy. During the physical exam, the participant will be asked questions about their general health, questions about any problems that they may be experiencing, and any medications they are taking.
* Blood tests: The participant will have blood drawn on the first and fifteenth days of the first three months of therapy. After that, the participant will have blood drawn every month for the remainder of the first year of treatment and the every other month until the end of therapy. These tests will be used to determine if the participant is having any side effects related to the study drug.
* Electrocardiograms (EKG): The participant will have an EKG performed on the first day of the first three months of therapy. After that, the participant will have an EKG every other month until the end of the first year of therapy. After the first year of therapy, the participant will have an EKG every 3 months during the second year of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed hormone receptor positive (HR+) HER2 negative stage II (except T2N0) or stage III invasive breast cancer. Evaluation for metastatic disease is not required in the absence of symptoms.
* Men and both pre- and postmenopausal women are eligible.
* Prior Treatment:

  * Participants may have received (neo)adjuvant chemotherapy, but must be at least 30 days after last dose, with no more than grade 1 residual toxicity at time of screening.
  * Participants may have received adjuvant radiotherapy, but must be at least 30 days after last dose , with no more than grade 1 residual toxicity at the time of screening.
  * If most recent therapy was surgery, participants must be at least 30 days out from definitive surgery with no active wound healing complications.
* Participants must have demonstrated ability to tolerate endocrine therapy by prior successful completion of at least 1 month of tamoxifen or aromatase inhibitor (AI) therapy without significant adverse events, and in the opinion of the treating physician any ongoing toxicity does not preclude ability to continue on tamoxifen or AI for at least a projected 2 year continuous duration. Ongoing use of any endocrine therapy, including tamoxifen, letrozole, anastrozole, or exemestane, is allowed. Patients may enroll within 2 years of beginning endocrine therapy, as long as there is a plan for at least 2 more years of adjuvant endocrine therapy.
* ECOG performance status 0-1
* Age ≥18 years.
* Normal organ and marrow function
* Baseline QTc ≤ 480 ms
* The effects of palbociclib on the developing human fetus are unknown. Women who might become pregnant must use adequate contraception
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Concurrent therapy with other investigational agents.
* Prior therapy with any CDK4/6 inhibitor.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A isoenzymes are ineligible.
* Current use of drugs that are known to prolong the QT interval
* Subjects with organ allograft requiring immunosuppression.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study. Breastfeeding should be discontinued prior to entry onto the study.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: ductal carcinoma in situ of the breast, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* No ongoing combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-01; Primary Completion 2018-05 (Actual); Study Completion 2024-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Mayer, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (10):
- United States (10):
  - University of California, San Francisco, San Francisco, California
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - MGH/North Shore Cancer Center, Danvers, Massachusetts
  - DF/DWCC at Milford Regional Cancer Center, Milford, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire
  - University of Pennsylvania-Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mayer EL, DeMichele A, Rugo HS, Miller K, Waks AG, Come SE, Mulvey T, Jeselsohn R, Overmoyer B, Guo H, Barry WT, Huang Bartlett C, Koehler M, Winer EP, Burstein HJ. A phase II feasibility study of palbociclib in combination with adjuvant endocrine therapy for hormone receptor-positive invasive breast carcinoma. Ann Oncol. 2019 Sep 1;30(9):1514-1520. doi: 10.1093/annonc/mdz198. PMID 31250880

RESULTS

PARTICIPANT FLOW:
Groups:
- Palbociclib With Adjuvant Endocrine Therapy: Palbociclib: 125 mg PO qd 21 days on, 7 days off Endocrine Therapy: Tamoxifen 20mg, Letrozole 2.5mg, Anastrozole 1mg, or Exemestane 25mg PO qd
Period: Overall Study
Arm/Group | Palbociclib With Adjuvant Endocrine Therapy
Started | 162
Treatment Discontinuation Evaluable | 152 (Evaluable population excludes participants who discontinue early for reasons unrelated to treatment.)
Completed | 102
Not Completed | 60
Not completed — Adverse Event | 14
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 31
Not completed — patient non-compliance | 3
Not completed — Lost to Follow-up | 2
Not completed — recurrence | 4
Not completed — ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Palbociclib With Adjuvant Endocrine Therapy
Number analyzed (Participants) | 162
Age, Customized [Count of Participants; unit: Participants]
  Age, <50 years | 69
  Age, >50 years | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 144
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 162
Type of prior neo/adjuvant chemotherapy [Count of Participants; unit: Participants]
  None | 33
  Neoadjuvant | 60
  Adjuvant | 63
  Both | 4
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: 2-Year Treatment Discontinuation Rate
Description: The 2-year treatment discontinuation rate is the percentage of participants who do not complete the palbociclib treatment per protocol for reasons due to toxicity, withdrawal of consent to be treated, or other events related to tolerability in uncensored participants. Participants who discontinued palbociclib early for reasons that were not treatment-related were censored.
Time Frame: Evaluate upon completion of palbociclib, up to 2 years of treatment completion.
Population: The analysis population is comprised of all uncensored participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib With Adjuvant Endocrine Therapy
Number analyzed (Participants) | 152
percentage of participants | 31 [24 to 39]
Statistical Analysis 1: Comparison: Palbociclib With Adjuvant Endocrine Therapy; Primary objective is treatment discontinuation rate at 2 yr for patients receiving Palbociclib therapy. If the true rate of discontinuation by two years is 48% or higher, treatment duration will be considered not feasible and not worthy of further study. If the rate of discontinuation is 33.3% or less, the 2 yr duration will be deemed feasible and worthy of further study. Using a one-sided alpha = 0.025, there is > 90% power to reject the null hypothesis in favor of feasibility; Test type: Other — Exact binomial test; p = 0.0011, Exact binomial test

2. Secondary Outcome: 2-year Treatment Discontinuation Rate by Aromatase Inhibitor and Tamoxifen-based Therapy Subgroup
Description: The 2-year treatment discontinuation rate is the percentage of participants who do not complete the palbociclib treatment per protocol for reason due to toxicity, withdrawal of consent to be treated, or other events related to tolerability of all enrolled participants.
Time Frame: Evaluate upon completion of palbociclib, up to 2 years of treatment completion.
Population: The analysis population is comprised of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Aromatase Inhibitor + Palbociclib: participants who received an Aromatase inhibitor as their endocrine therapy with Palbociclib
- Tamoxifen + Palbociclib: participants who received Tamoxifen as their endocrine therapy with Palbociclib
Arm/Group | Aromatase Inhibitor + Palbociclib | Tamoxifen + Palbociclib
Number analyzed (Participants) | 102 | 60
percentage of participants | 28 [20 to 38] | 35 [23 to 48]

3. Secondary Outcome: Grade 3-4 Treatment-Related Neutropenia Toxicity Rate
Description: Grade 3-4 treatment-related neutropenia toxicity rate is the percentage of participants experiencing at least one grade 3-4 neutropenia AE with treatment attribution of possible, probable or definite based on NCI Common Toxicity Criteria for Adverse Events version 4 (CTCAEv4) during the time of observation on treatment as reported on case report forms.
Time Frame: AE data collected every cycle from the time of the first dose of study treatment, through the study and until 30 days after removal from study or death, whichever occurs first. Therefore, AEs were observed up to 2 years plus 30 days.
Population: The analysis population is comprised of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib With Adjuvant Endocrine Therapy
Number analyzed (Participants) | 162
percentage of participants | 54 [46 to 62]

4. Secondary Outcome: All Grade Treatment-Related Fatigue Toxicity Rate
Description: All grade treatment-related fatigue toxicity rate is the percentage of participants experiencing at least one grade 1-4 fatigue AE with treatment attribution of possible, probable or definite based on NCI Common Toxicity Criteria for Adverse Events version 4 (CTCAEv4) during the time of observation on treatment as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population is comprised of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib With Adjuvant Endocrine Therapy
Number analyzed (Participants) | 162
percentage of participants | 76 [69 to 82]

5. Secondary Outcome: All GradeTreatment-Related Alopecia Toxicity Rate
Description: All grade treatment-related alopecia toxicity rate is the percentage of participants experiencing at least one grade 1-4 alopecia AE with treatment attribution of possible, probable or definite based on NCI Common Toxicity Criteria for Adverse Events version 4 (CTCAEv4) during the time of observation on treatment as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population is comprised of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib With Adjuvant Endocrine Therapy
Number analyzed (Participants) | 162
percentage of participants | 28 [22 to 36]

6. Post Hoc Outcome: Rate of Treatment Related Discontinuation
Description: The 2-year treatment discontinuation rate is the percentage of participants who do not complete the palbociclib treatment per protocol for reasons due to toxicity, withdrawal of consent to be treated, or other events related to tolerability in all enrolled participants.
Time Frame: Evaluate upon completion of combination therapy with endocrine therapy plus palbociclib, up to 2 years of treatment completion.
Population: The analysis population is comprised of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib With Adjuvant Endocrine Therapy
Number analyzed (Participants) | 162
percentage of participants | 63 [55 to 70]

ADVERSE EVENTS:
Time Frame: AE data collected every cycle from the time of the first dose of study treatment, through the study and until 30 days after removal from study or death, whichever occurs first. Therefore, AEs were observed up to 2 years plus 30 days.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Palbociclib With Adjuvant Endocrine Therapy
All-Cause Mortality (participants affected / at risk) | 0/162
Serious Adverse Events (participants affected / at risk) | 96/162
Other Adverse Events (participants affected / at risk) | 162/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib With Adjuvant Endocrine Therapy (N=162)
Cardiac disorders - Other, specify (Cardiac disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Breast infection (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 78
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib With Adjuvant Endocrine Therapy (N=162)
Anemia (Blood and lymphatic system disorders) | 42
Lymph node pain (Blood and lymphatic system disorders) | 2
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Chest pain - cardiac (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 7
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 4
Vertigo (Ear and labyrinth disorders) | 2
Vestibular disorder (Ear and labyrinth disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Chills (General disorders) | 3
Edema limbs (General disorders) | 9
Fatigue (General disorders) | 58
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Localized edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 4
Bronchial infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT02040857/Prot_SAP_000.pdf